CLINICAL TRIAL: NCT07322328
Title: Effects of Hypo-pressive Exercises and Pelvic Floor Muscle Training on the Severity of Stress Urinary Incontinence and Quality of Life in Postpartum Women
Brief Title: Effect of Hypo-pressive Exercises and Pelvic Floor Muscle Training in Postpartum Stress Urinary Incontinence Women
Acronym: SUI PFMT HE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Principal Investigator, Dr. Mehwish Khalid, Assistant Professor, Lahore University of Biological and Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DPT/ERB/29; U1111-1332-3272 (Registry Identifier: Isma Habib)
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Stress Urinary Incontinence (SUI); Stress Urinary Incontinence in Women
Keywords: Post-partum stress urinary incontinence; Hypopressive exercises; Pelvic floor muscle training; Quality of life
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypopressive Exercises (Experimental): Hypo-pressive Exercise (HE) training involves ribcage expansion and apnea to generate negative pressure, which in turn activates the deep core and pelvic floor muscles instinctively. Activating type I muscle fibers improves postural control, endurance, and coordination.
  Interventions: Other: hypo-pressive exercise
- Pelvic Floor Muscle Training (Active Comparator): Pelvic Floor Muscle Training (PFMT) through voluntary contraction and resistance training strengthens pelvic floor musculature. In addition, these exercises have the potential to improve control over urine and fecal incontinence.
  Interventions: Other: pelvic floor muscle training

INTERVENTIONS:
Other: hypo-pressive exercise — Exercise is performed 3 times per week for 6 weeks with moderate intensity for 20 min/session which includes diaphragmatic breathing, apnea, postural alignment (standing, seated, kneeling), and pelvic floor co-activation).
  Arms: Hypopressive Exercises
Other: pelvic floor muscle training — Exercise is performed 3 times per week for 6 weeks with submaximal voluntary contraction (include both slow holds and quick flicks) for 20 min/session (each session includes multiple sets of 8 repetitions, hold for 5 seconds, with rest intervals). These Kegel exercises are performed in different positions.
  Arms: Pelvic Floor Muscle Training

SUMMARY:
Postpartum stress urinary incontinence is a widespread condition characterized by involuntary loss of urine during physical exertion, such as sneezing, coughing, or lifting heavy weights. Most frequently occur in multiparous women with vaginal delivery, who are obese, constipated, or with low maternal education. Damage to the levator ani muscle complex and adjacent fascia during childbirth affects urethral mobility and consequently results in sphincter insufficiency.

Hypopressive exercises involve breathing techniques that regulate the intra-abdominal pressure. HE has been recently recognized for benefits such as pelvic floor muscle (PFM) strength, endurance, postural control, core muscle activation, and respiratory capacity, which efficiently improve symptom severity and quality of life in postpartum women.

Pelvic floor muscle training (PFMT) is a set of frequent voluntary contractions designed to improve strength, coordination, and control. PFMT is considered as standard treatment protocol for urinary incontinence and other postpartum complications.

The International Consultation on Incontinence Questionnaire-Short Form (ICIQ-UI-SF) and the Incontinence Quality of Life (IQOL) are used to assess symptom severity and quality of life, respectively. This study seeks to bridge that gap by evaluating and comparing the outcomes of HE and PFMT in postpartum women experiencing SUI. This research aims to support postpartum recovery, improve women's daily functioning, and enhance their overall well-being.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 20 and 40 years old
* Multiparous women
* Postpartum women ≤ 6 months.
* Vaginal deliveries.
* Women diagnosed with stress urinary incontinence within 6 weeks to six months

Exclusion Criteria:

* Neurological disorder
* Metabolic issue
* Abdominal and pelvic surgery in previous years
* Mentally retarded
* Pregnant women

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — postpartum women
Enrollment: 38 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2026-05-22 (Estimated); Study Completion 2026-05-22 (Estimated)

PRIMARY OUTCOMES:
Symptoms severity | 6 weeks
  Symptom severity due to SUI will assessed by International Consultation on Incontinence Questionnaire Urinary Incontinence short form (ICIQUI-SF) is a standardized, validated, self-administered questionnaire used to assess the severity of urinary incontinence (UI), influence quality of life, and situational triggers of leakage. It consists of four items: frequency of urine leakage, amount of urine leakage, overall impact of UI on daily life (rated on a 0-10 scale), and a self-diagnostic item asking when urine leaks (non-scored). The ICIQ-UI-SF showed a Cronbach's alpha value from 0.7 to 0.8, representing good internal consistency

SECONDARY OUTCOMES:
Incontinence Quality of life | 6 weeks
  Incontinence Quality of life (I-QOL) is a self-assessment tool that is repeatedly utilized in people with UI. The 22-item I-QOL has three subscales: social embarrassment (SE), psychosocial impact (PSI), and avoidance and limiting behaviors (ALB). It based on Likert scale which comprises of five point, i.e. 1=always, 2=often, 3=sometimes, 4=rarely and 5=never. The IQOL showed a Cronbach's alpha value was 0.96, representing good internal consistency.

CONTACTS AND LOCATIONS:
Locations (1):
- Lahore University of Biological and Applied Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
After the publication of the research
Supporting Information: Study Protocol
Time Frame: July 2026- till any update